CLINICAL TRIAL: NCT06962566
Title: Effects of Exercise at Different Times of Day on 72-hour Eating Behaviours and Physical Activity in Physically Inactive Adults
Brief Title: Effects of Different Timing of Brisk Walking on Human Behaviours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yung-Chih Chen, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202405HM084-1
Record Dates: First submitted 2025-04-23; First posted 2025-05-08 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Physical Activity; Energy Intake; Sedentary Behavior
Keywords: Timing of exercise; Morning exercise; Evening exercise; Behavioural compensation
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning exercise (Experimental): Brisk walking in the morning
  Interventions: Behavioral: Morning exercise
- Evening exercise (Experimental): Brisk walking in the evening
  Interventions: Behavioral: Evening exercise

INTERVENTIONS:
Behavioral: Morning exercise — Participants performed a 45-minute treadmill brisk walking in the morning between 08:00 to 11:00 AM.
  Arms: Morning exercise
Behavioral: Evening exercise — Participants performed a 45-minute treadmill brisk walking in the evening between 18:00 to 21:00 PM.
  Arms: Evening exercise

SUMMARY:
The purpose of this project is to investigate the effects of exercise at different times of day on 72-hour eating behaviour, physical activity and sedentary behaviour in physically inactive adults.

DETAILED DESCRIPTION:
Eligibility and Consent Confirmation Prior to the one-week preliminary test, participants underwent eligibility screening, including measurements of height, weight, and body composition. After the researchers provided a detailed explanation of the experimental procedures, participants decided whether to participate in the study. Eligible participants then completed a 10-minute treadmill walking session (6.4 km/h for males and 6.0 km/h for females) to familiarize themselves with the exercise intensity. Subsequently, the researchers explained the use of pedometers and distributed dietary record forms.

During a one-week preliminary test, participants were instructed to record their physical activity levels measured in steps, sleep duration including wake-up and sleep times, and dietary behaviours through photographs taken (2 weekdays and 1 weekend day) over a period of 7 consecutive days. Participants were allowed to take part in this study, once they met the inclusion criteria: 1) an average daily step count of less than 7,500 over the course of the week and 2) a wake-up time no later than 11:00 AM).

Exercise intervention During the main trials, two main trials, separated by at least one week, were conducted - exercise in the morning (08:00 to 11:00 AM) or exercise in the evening (18:00 to 21:00 PM).

In both trials, participants completed the first Visual Analogue Scale (VAS) for subjective appetite upon waking, wore a pedometer and an accelerometer, and recorded energy intake and physical activity over a 3-day period (the day before exercise intervention, the exercise day and the day after exercise intervention). Upon arrival at the laboratory, participants completed the second VAS, followed by a 15-minute waiting period before commencing the exercise. Participants then performed a 45-minute treadmill brisk walk (6.4 km/h for males, 6.0 km/h for females), followed by a 15-minute rest period, after which they completed the third VAS.

Heart rate and Rating of Perceived Exertion (RPE) were measured every 15 minutes during exercise. Energy balance (e.g., energy intake and spontaneous physical activity) was assessed using a food diary, Actigraph wGT3x-BT accelerometer (Actigraph Co., Ltd., Pensacola, FL, USA), and pedometer (Realalt, Goldhat Ltd., UK), which were worn starting from the night two days before the experiment and removed after waking up two days post-experiment.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 50 years, with a BMI ranging from 19 to 27 kg/m².
* Classified as having "low" physical activity levels (750 Metabolic Equivalents / week) according to the International Physical Activity Questionnaire (IPAQ).
* Engaged in moderate-intensity exercise for no more than 3 days per week and less than 30 minutes per session in the 3 months preceding the study.
* Maintained a stable body weight (± 3 kg) during the 3 months prior to the main experiment.
* Not taking any medications, supplements, or vitamins that might affect food intake, appetite, physical activity, weight loss, or metabolism.
* Free from cardiovascular and metabolic diseases.
* Not pregnant or planning to become pregnant.
* Not currently on a diet or undergoing any specific dietary interventions (e.g., intermittent fasting, ketogenic diet).
* No injuries or surgical wounds preventing physical activity.
* Regular sleep patterns, averaging 7-9 hours per night, with no shift work.
* No habits of heavy alcohol consumption or smoking.

Exclusion Criteria:

* Personal history of/existing diabetes, cardiovascular disease, metabolic disease or dyslipidaemia.
* Taking medications that may influence lipid or carbohydrate metabolism or immune system function.
* Unable to take part in exercise for any reason (e.g., injury or disability) or a positive response to any questions on the Physical Activity Readiness questionnaire (PAR-Q).

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Physical activity | 72 hours (24 hours before exercise day, exercise day and 24 hours after exercise day)
  Changes in physical activity intensity (minutes and percentage during 72 hours) and levels (minutes and percentage during 72 hours) between trials
Energy intake | 72 hours (24 hours before exercise day, exercise day and 24 hours after exercise day)
  Changes in total and macronutrient energy intake between trials
Sedentary behaviour | 72 hours (24 hours before exercise day, exercise day and 24 hours after exercise day)
  Changes in sedentary behaviour (minutes and percentage during 72 hours) between trials

SECONDARY OUTCOMES:
Heart Rate | During 45 minutes exercise
  Changes in heart rate (bpm) during exercise between trials
Rating of Perceived Exertion (RPE) | During 45 minutes exercise
  Changes in Rating of Perceived Exertion using Borg 6-20 scale (6 indicates no exertion and 20 indicates maximal effort) during exercise between trials
Visual analogue scale (VAS) | Baseline upon wake up in the morning,15 minutes before exercise and 15 minutes after exercise
  Changes in Visual analogue scale (appetite) using 0-100 mm scale (0 indicates not at all and 100 indicates very much) during exercise between trials

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan